CLINICAL TRIAL: NCT06216301
Title: LUNAR-2: Pivotal, Randomized, Open-Label Study of Tumor Treating Fields (TTFields, 150 kHz) Concomitant With Pembrolizumab and Platinum-based Chemotherapy for the Treatment of Metastatic Non-Small Cell Lung Cancer
Brief Title: LUNAR-2: TTFields With Pembrolizumab + Platinum-based Chemotherapy for Metastatic NSCLC
Acronym: LUNAR-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-44
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: NSCLC; Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — pembrolizumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm 1: NovoTTF-200T, Pembrolizumab, and Platinum-based Chemotherapy (Experimental): Subjects in this arm receive three treatments - TTFields using the NovoTTF-200T device, pembrolizumab, and platinum-based chemotherapy.
  Interventions: Device: NovoTTF-200T; Drug: Pembrolizumab; Drug: Platinum based chemotherapy
- Arm 2: Pembrolizumab and Platinum-based Chemotherapy (Active Comparator): Subjects in this arm receive two treatments - pembrolizumab and platinum-based chemotherapy.
  Interventions: Drug: Pembrolizumab; Drug: Platinum based chemotherapy

INTERVENTIONS:
Device: NovoTTF-200T — The NovoTTF-200T is a portable, battery operated system intended for continuous home use, which delivers TTFields at a frequency of 150kHz to the subject by means of insulated transducer arrays. TTFields physically disrupt the rapid cell division exhibited by cancer cells. The physical disruption induced by TTFields can lead to to downstream immunogenic cell death.
  Arms: Arm 1: NovoTTF-200T, Pembrolizumab, and Platinum-based Chemotherapy
Drug: Pembrolizumab — Pembrolizumab is an immune checkpoint inhibitor that helps the immune system recognize and attack cancer cells.
Drug: Platinum based chemotherapy — Platinum-based chemotherapy is a standard chemotherapy regimen commonly used in the treatment of non-small cell lung cancer

SUMMARY:
This study, known as LUNAR-2, aims to investigate the effectiveness and safety of using TTFields, delivered by the NovoTTF-200T device, concomitantly administered with pembrolizumab and platinum-based chemotherapy for patients with advanced non-small cell lung cancer that has spread to other parts of the body. The primary goals of the study are to assess overall survival and progression-free survival. Secondary objectives include analyzing outcomes based on the specific histology (subtype) of the lung cancer.

DETAILED DESCRIPTION:
LUNAR-2 is a pivotal, randomized, open-label study that aims to evaluate the effectiveness and safety of Tumor Treating Fields (TTFields) concomitantly administered with pembrolizumab and platinum-based chemotherapy for the treatment of metastatic non-small cell lung cancer (NSCLC).

The primary objectives of the study are to assess overall survival (OS) and progression-free survival (PFS) in subjects treated with TTFields, pembrolizumab, and platinum-based chemotherapy compared to those treated with pembrolizumab and platinum-based chemotherapy alone. PFS will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

The secondary endpoints of this study will evaluate PFS and OS, stratified by the specific histological subtype of NSCLC and PD-L1 Tumor Proportion Score (TPS).

The population will consist of subjects with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 and will be stratified as follow:

1. Histology - Squamous vs. non-squamous
2. PD-L1 expression level - TPS <1% vs. 1% ≤TPS <50% vs. TPS ≥50%
3. Prior treatment with immunotherapy - yes vs. no

The study will be conducted globally at approximately 130 participating sites. The study device, NovoTTF-200T, is a portable, battery-operated system that delivers TTFields at a frequency of 150kHz. It utilizes insulated transducer arrays to deliver electric forces intended to disrupt cancer cell division.

ELIGIBILITY:
Inclusion Criteria

* ≥22 years of age in the USA

  ≥18 years of age outside of the USA.
* Histologically or cytologically diagnosis of stage 4 (according to Version 8 of the American Joint Committee on Cancer [AJCC] criteria) non-squamous or squamous NSCLC.
* Evaluable (measurable or non-measurable) disease in the thorax per RECIST v1.1.
* Have not received prior systemic treatment for their metastatic NSCLC. Subjects who received adjuvant, neoadjuvant chemotherapy or chemoradiotherapy with curative intent for non-metastatic disease are eligible if the therapy was completed at least 12 months prior to the development of metastatic disease.
* ECOG Performance Status (PS) of 0-1.
* Adequate hematologic and end-organ function

  o For subjects not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN (unless participant is receiving anticoagulant therapy as long as INR or aPTT is within therapeutic range of intended use of anticoagulants).
* A female participant is eligible to participate if she is not pregnant, not breastfeeding
* If male subject with a female partner(s) of child-bearing potential, must agree to use an effective contraception
* All subjects must sign written informed consent.

Exclusion Criteria:

All individuals meeting any of the following exclusion criteria will be excluded from study participation:

* Mixed small cell and NSCLC histology.
* EGFR sensitizing mutation and/or ALK translocation, and/or ROS1 and/or RET targetable gene rearrangement, and/or METex14 skipping mutation, and/or NTRK1/2 gene fusion and/or BRAF V600 mutations directed therapy is indicated or planned for other targeted therapy, where such testing and therapy is locally approved and available.
* Has received systemic therapy for metastatic disease.
* Had major surgery <3 weeks prior to randomization
* Received radiation therapy to the lung that is > 30 Gy within 6 months of randomization.
* Has received prior radiotherapy within 2 weeks of randomization. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Is expected to require any other form of antineoplastic therapy while on study.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

  * Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has symptomatic Central Nervous System (CNS) metastases and/or carcinomatous meningitis. Subjects with asymptomatic CNS metastases or with previously treated brain metastases may participate provided they were treated before randomization (if applicable) and are neurologically stable and without requirement of steroid treatment for at least 7 days prior to randomization.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior randomization. Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
* Had prior treatment with any other anti-PD-1, or PD-L1 or PD-L2 agent or an antibody or a small molecule targeting other immuno-regulatory receptors or mechanisms in the 12 months prior to randomization.
* Participation in another clinical study with an investigational agent or device during the 4 weeks prior to randomization.
* Concurrent treatment with other experimental treatments for NSCLC while in the study.
* Has a known sensitivity to any component of the planned systemic therapies (pembrolizumab, cisplatin/carboplatin, pemetrexed/paclitaxel/nab-paclitaxel) .
* Pregnant or breastfeeding
* Admitted to an institution by administrative or court order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 6 years
  To compare OS in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy compared to OS of those treated with pembrolizumab and platinum-based chemotherapy alone (superiority analysis).
Progression Free Survival (PFS) | up to 6 years
  To compare PFS per RECIST v1.1 as assessed by BICR, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy compared to PFS of those treated with pembrolizumab and platinum-based chemotherapy alone (superiority analysis)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 6 years
  Progression Free Survival (PFS) per RECIST v1.1 as assessed by BICR, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone according to histology.
Overall Survival (OS) | up to 6 years
  Overall Survival (OS) in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone according to histology.
Progression Free Survival (PFS) | up to 6 years
  PFS per RECIST v1.1 as assessed by BICR, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone according to PD-L1 Tumor Proportion Score (TPS).
Overall Survival (OS) | up to 6 years
  OS in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone according to PD-L1 TPS.
Progression Free Survival (PFS) | up to 6 years
  PFS per RECIST v1.1 as assessed by BICR at 6 (PFS6), 12 (PFS12), 24 (PFS24), and 36 (PFS36) months in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
1, 2, and 3-year Survival Rate | up to 6 years
  1-, 2- and 3-year survival rate in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Objective Response Rate (ORR) | up to 6 years
  Objective Response Rate (ORR) per RECIST v1.1 as assessed by BICR, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Duration of Response (DoR) | up to 6 years
  Duration of Response (DoR) per RECIST v1.1 as assessed by BICR, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Disease Control Rate (DCR) | up to 6 years
  Disease Control Rate (DCR) per RECIST v1.1 as assessed by BICR, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Progression Free Survival (PFS) | up to 6 years
  PFS per RECIST v1.1 as assessed by the investigator, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Objective Response Rate (ORR) | up to 6 years
  ORR per RECIST v1.1 as assessed by the investigator, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Duration of Response (DoR) | up to 6 years
  DoR per RECIST v1.1 as assessed by the investigator, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Disease Control Rate (DCR) | up to 6 years
  DCR per RECIST v1.1 as assessed by the investigator, in subjects treated with TTFields concomitant with pembrolizumab and platinum-based chemotherapy and of those treated with pembrolizumab and platinum-based chemotherapy alone.
Adverse Events | up to 6 years
  Toxicity profile of TTFields concomitant with pembrolizumab and platinum-based chemotherapy. The analyses will be performed based on the incidence, severity, frequency of adverse events, and their association with study treatments.

CONTACTS AND LOCATIONS:
Locations (90):
- United States (35):
  - Central Alabama Research, Birmingham, Alabama
  - Western Regional Medical Center, LLC, Goodyear, Arizona
  - St. Jude Herritage Medical Group, Fullerton, California
  - Hoag Family Cancer Institute - Hoag Memorial Hospital, Newport Beach, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Florida Cancer Affiliates - Ocala Oncology, Ocala, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwest Oncology & Hematology, Barrington, Illinois
  - Elmhurst Hospital Nancy Knowles Cancer Center, Elmhurst, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Cancer Treatment Centers of America (CTCA), Zion, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Luminis Health Radiation Oncology - Anne Arundel Health System, Annapolis, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center - Overland Park, Overland, Missouri
  - New York Cancer & Blood Specialists (NYCBS), New Hyde Park, New York
  - New York Cancer & Blood Specialists (NYCBS), New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - New York Cancer & Blood Specialists (NYCBS), Shirley, New York
  - New York Cancer & Blood Specialists (NYCBS), The Bronx, New York
  - WakeMed Health & Hospitals, Cary, North Carolina
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - AHN Cancer Center, Pittsburgh, Pennsylvania
  - Old Parkland Hospital Hematology Oncology Clinic, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - DHR Health Oncology Institute, Edinburg, Texas
  - Methodist Richardson Cancer Center, Richardson, Texas
  - Jason Bates at University of Texas Health Science Center, San Antonio, Texas
  - MultiCare Regional Cancer Center, Auburn, Washington
  - MultiCare Regional Cancer Center, Gig Harbor, Washington
  - MultiCare Regional Cancer Center, Puyallup, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Austria (3):
  - Universitaetsklinik fuer Innere Medizin V Innsbruck, Innsbruck
  - University Hospital Salzburg, Salzburg
  - Karl Landsteiner Institut fur Lungenforschung und pneumologische Onkologie c/o Klinik Floridsdorf, Vienna
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - AZ Maria Middelares - Campus Maria Middelares, Ghent
- Czechia (3):
  - Fakultni nemocnice Olomouc FNOL, Olomouc
  - Nemocnice Agel Ostrava-Vitkovice / Agel Ostrava-Vitkovice Hospital, Ostrava
  - General University Hospital in Prague, Prague
- France (8):
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - CHU Limoges, Limoges
  - Hopital Europeen, Marseille
  - Hopital Prive du Confluent, Nantes
  - Institut Curie, Paris
  - CHU de Bordeaux, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Nouvel Hopital Civil (NHC), Strasbourg
- Germany (6):
  - Evangelische Lungenklinik Berlin, Berlin
  - University Hospital Giessen, ZIM IV, Giessen
  - Krankenhaus Martha-Maria Halle-Dolau, Halle
  - Thoraxklinik Heidelberg, Heidelberg
  - Klinik Loewenstein gGmbH, Löwenstein
  - Pius-Hospital Oldenburg, Oldenburg
- Hungary (3):
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
- Israel (2):
  - Emek Medical Center, Afula
  - Bnai zion MC, Haifa
- Italy (8):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria
  - Humanitas Gavazzeni, Bergamo
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Ferrara
  - IRCCS - Istituto Romagnolo per lo Studio Dei Tumori, Dino Amadori, Meldola
  - Azienda Sanitaria Territoriale Pesaro Urbino, Pesaro
  - Universita Campus Bio-Medico di Roma (UCBM) - Policlinico Universitario, Roma
  - Ospedale Isola Tiberina Gemelli, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
- Netherlands (4):
  - Rijnstate Ziekenhuis, Arnhem
  - Medisch Centrum Leeuwarden (MCL) - Oncologisch Centrum Leeuwarden (OCL), Friesland
  - St. Jansdal ziekenhuis, Harderwijk
  - St Antonius Ziekenhuis, Utrecht
- Uniwersytecki Szpital Kliniczny, Poznan, Poland
- Singapore (3):
  - NCCS Singapore, Singapore
  - Curie Oncology, Singapore
  - Icon Cancer Centre Singapore (Singapore Oncology Consultants), Singapore
- Spain (10):
  - Hospital Universitario del Vinalopo, Elche, Alicante
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Clinica Mi Tres Torres Barcelona - Giromed Institute, Barcelona, Catalonia
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Clinica Universidad de Navarra (Madrid), Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
- Switzerland (2):
  - Cantonal Hospital Baden, Baden
  - HFR Freiburg-Kantonsspital, Fribourg

IPD SHARING:
Plan to Share IPD: No